CLINICAL TRIAL: NCT05175105
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Mitapivat in Pediatric Subjects With Pyruvate Kinase Deficiency Who Are Not Regularly Transfused, Followed by a 5-Year Open-label Extension Period
Brief Title: A Study to Evaluate the Efficacy and Safety of Mitapivat in Pediatric Participants With Pyruvate Kinase Deficiency (PKD) Who Are Not Regularly Transfused, Followed by a 5-Year Extension Period
Acronym: ACTIVATE-Kids
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG348-C-023; 2021-003333-11 (EudraCT Number)
Record Dates: First submitted 2021-11-22; First posted 2022-01-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Pyruvate Kinase Deficiency; Pediatric Hemolytic Anemia
Keywords: Anemia; Hematologic Diseases; Metabolic Diseases; Mitapivat; AG-348; ACTIVATE-Kids; PK Deficiency
MeSH Terms: conditions — Anemia; Hematologic Diseases; Metabolic Diseases; Pyruvate Kinase Deficiency of Red Cells | interventions — mitapivat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mitapivat (Experimental): Double-Blind Period: Participants will receive mitapivat orally, at doses based on age and weight, for 8 weeks in the dose titration period and for 12 weeks in the fixed-dose period.
  Interventions: Drug: Mitapivat
- Placebo (Placebo Comparator): Double-Blind Period: Participants will receive mitapivat-matching placebo orally for 8 weeks in the dose titration period and for 12 weeks in the fixed-dose period.
  Interventions: Drug: Mitapivat-matching placebo
- Mitapivat (OLE period) (Experimental): Participants who have completed the double-blind period will be eligible to receive mitapivat for up to 5 years in the OLE period. Participants entering the OLE period will first receive blinded mitapivat and placebo for 8 weeks to maintain the double-blind treatment assignment before being transitioned to only receive active, open-label drug (mitapivat).
  Interventions: Drug: Mitapivat; Drug: Mitapivat-matching placebo

INTERVENTIONS:
Drug: Mitapivat — Tablets or granules
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate
  Arms: Mitapivat; Mitapivat (OLE period)
Drug: Mitapivat-matching placebo — Tablets or granules
  Arms: Mitapivat (OLE period); Placebo

SUMMARY:
Study ACTIVATE-Kids (AG348-C-023) will evaluate the efficacy and safety of orally administered mitapivat as compared with placebo in pediatric participants with pyruvate kinase deficiency (PKD) who are not regularly receiving blood transfusions. Participants will be randomized 2:1 to receive either mitapivat or matching placebo. Randomization will be stratified by age (1 to < 6 years, 6 to < 12 years, 12 to < 18 years). Participants will be dosed by age and weight during a double-blind period consisting of an 8-week dose titration period followed by a 12-week fixed-dose period. Participants who complete the double-blind period will be eligible to receive mitapivat for up to 5 years in the open-label extension (OLE) period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the participant, or the participant's legally authorized representative, parent(s), or legal guardian, and the participant's assent, where applicable (informed consent/assent) must be obtained before any study-related procedures are conducted, and participants must be willing to comply with all study procedures for the duration of the study;
* Aged 1 to <18 years. Participants between 12 and 24 months of age must weigh a minimum of 7 kilograms (kg);
* Clinical laboratory confirmation of pyruvate kinase deficiency (PKD), defined as documented presence of at least 2 mutant alleles in the pyruvate kinase L/R (PKLR) gene, of which at least 1 is a missense mutation, as determined per the genotyping performed by the study central genotyping laboratory;
* No more than 5 red blood cell (RBC) transfusions in the 52-week period before providing informed consent/assent and no RBC transfusions ≤12 weeks before administration of the first dose of study drug;
* Hemoglobin concentration ≤10 grams per deciliter (g/dL) for participants 12 to <18 years of age or ≤9 g/dL for participants 1 to <12 years of age during the screening period. Hb concentration must be based on an average of at least 2 Hb concentration measurements (separated by ≥7 days) collected during the screening period;
* Receiving folic acid supplementation as part of routine clinical care for at least 21 days before administration of the first dose of study drug, to be continued during study participation;
* Female participants who have attained menarche and/or breast development in Tanner Stage 2 must be abstinent of sexual activities that may induce pregnancy as part of their usual lifestyle, or agree to use 2 forms of contraception, 1 of which must be considered highly effective, from the time of informed consent/assent, throughout the study, and for 28 days after the last dose of study drug (including the time required to dose taper). The second form of contraception can include an acceptable barrier method.

Exclusion Criteria:

* Pregnant or breastfeeding;
* Homozygous for the R479H mutation or have 2 nonmissense mutations, without the presence of another missense mutation, in the PKLR gene as determined per the genotyping performed by the study central genotyping laboratory;
* History of malignancy;
* History of active and/or uncontrolled cardiac or pulmonary disease or clinically relevant QT prolongation within 6 months before providing informed consent/assent;
* Hepatobiliary disorders including, but not limited to:

  * Liver disease with histopathological evidence of cirrhosis or severe fibrosis;
  * Clinically symptomatic cholelithiasis or cholecystitis (participants with prior cholecystectomy are eligible);
  * History of drug-induced cholestatic hepatitis;
  * Aspartate aminotransferase >2.5×upper limit of normal (ULN) (unless due to hemolysis and/or hepatic iron deposition) and alanine aminotransferase >2.5×ULN (unless due to hepatic iron deposition);
* Renal dysfunction as defined by an estimated glomerular filtration rate <60 milliliters per minute (mL/min)/1.73 m^2;
* Nonfasting triglycerides >440 milligrams per deciliter (mg/dL) (5 millimoles per liter [mmol/L]);
* Active uncontrolled infection requiring systemic antimicrobial therapy;
* Participants with known active hepatitis B or hepatitis C virus infection;
* Participants with known human immunodeficiency virus (HIV) infection;
* History of major surgery (including splenectomy) ≤6 months before providing informed consent/assent and/or planning on undergoing a major surgical procedure during the screening or double-blind period;
* Current enrollment or past participation (within 90 days before the first dose of study drug or a time frame equivalent to 5 half-lives of the investigational study drug, whichever is longer) in any other clinical study involving an investigational study drug or device;
* Prior exposure to gene therapy, or bone marrow or stem cell transplantation;
* Currently receiving hematopoietic stimulating agents; the last dose must have been administered at least 28 days or a time frame equivalent to 5 half-lives (whichever is longer) before randomization;
* Receiving products that are strong inhibitors of CYP3A4/5 that have not been stopped for ≥5 days or a time frame equivalent to 5 half-lives (whichever is longer), or strong inducers of CYP3A4 that have not been stopped for ≥28 days or a time frame equivalent to 5 half-lives (whichever is longer), before randomization;
* Receiving anabolic steroids, including testosterone preparations, that have not been stopped for at least 28 days before randomization;
* Known allergy, or other contraindication, to mitapivat or its excipients (microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, mannitol, Opadry® II Blue [hypromellose, titanium dioxide, lactose monohydrate, triacetin, and Food, Drug, and Cosmetics blue dye number 2 (FD&C Blue #2)], Opadry® II White [hypromellose, titanium dioxide, lactose monohydrate, and triacetin], and magnesium stearate);
* Any medical, hematologic, psychological, or behavioral condition(s) or prior or current therapy that, in the opinion of the Investigator, may confer an unacceptable risk to participating in the study and/or could confound the interpretation of the study data; also included are:

  * Participants who are institutionalized by regulatory or court order.
  * Participants with any condition(s) that could create undue influence (including but not limited to incarceration, involuntary psychiatric confinement, and financial or familial affiliation with the Investigator or Sponsor).
* Receiving a pyruvate kinase activator that has not been stopped for ≥52 weeks before providing informed consent/assent.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving a Hemoglobin (Hb) Response | Baseline up to Week 20
  Hb response is defined as a ≥1.5 grams per deciliter (g/dL) (0.93 millimoles per liter [mmol/L]) increase in Hb concentration from baseline that is sustained at 2 or more scheduled assessments at Weeks 12, 16, and 20 during the double-blind period. The individual participant's baseline Hb concentration is defined as the average of all available Hb concentrations collected for that participant during the screening period up to the first dose of study drug.

SECONDARY OUTCOMES:
Average Change From Baseline in Hb Concentration at Weeks 12, 16, and 20 | Baseline, Weeks 12, 16, and 20
Maximal Change in Hb Concentration From Baseline During the Double-blind Period | Baseline up to Week 20
Change From Baseline in Estradiol Concentration | Baseline up to Week 286
Change From Baseline in Estrone Concentration | Baseline up to Week 286
Change From Baseline in Total Testosterone Concentration | Baseline up to Week 286
Change From Baseline in Free Testosterone Concentration in Participants ≥7 Years of Age or Tanner Stage ≥2 (Whichever Occurs First) | Baseline up to Week 286
Change From Baseline in Luteinizing Hormone Concentration in Participants ≥6 Years of Age | Baseline up to Week 286
Change From Baseline in Sexual Maturity Rating with Tanner Stage | Baseline up to Week 286
  Tanner Stage 1 corresponds to the prepubertal form, with progression to Tanner Stage 5, the final adult form.
Number of Female Participants With Development of Ovarian Cysts | Baseline up to Week 286
Change From Baseline in the Size of Ovarian Cysts in Female Participants | Baseline up to Week 286
Change From Baseline in Height-for-age Z-score | Baseline up to Week 286
Change From Baseline in Weight-for-age Z-score | Baseline up to Week 286
Change From Baseline in Body Mass Index (BMI)-for-age Z-score | Baseline up to Week 286
Change From Baseline in Bone Mineral Density (BMD) Z-score | Baseline up to Week 286
Average Change From Baseline in Indirect Bilirubin Concentration at Weeks 12, 16, and 20 | Baseline, Weeks 12, 16, and 20
Average Change From Baseline in Lactose Dehydrogenase (LDH) Concentration at Weeks 12, 16, and 20 | Baseline, Weeks 12, 16, and 20
Change From Baseline in Haptoglobin Concentration at Week 16 | Baseline, Week 16
Change From Baseline in Reticulocytes | Baseline up to Week 286
Change From Baseline in Serum Iron Concentration | Baseline up to Week 280
Change From Baseline in Serum Ferritin Concentration | Baseline up to Week 280
Change From Baseline in Total Iron-binding Capacity | Baseline up to Week 280
Change From Baseline in Transferrin/Transferrin Saturation | Baseline up to Week 280
Change from Baseline in Pediatric Quality of Life (PedsQL) Multidimensional Fatigue Scale | Baseline up to Week 280
  The PedsQL multidimensional fatigue scale yields a total score from age-appropriate validated questionnaire that asks for perceived fatigue within the domains of 'General', 'Sleep/Rest' and 'Cognitive'. Each domain consists of 6 questions that are rated from 0 to 4 (therefore total score can range from 0 to 72). A higher total score indicates greater fatigue (i.e., worse outcome).
Change from Baseline in PedsQL Generic Core Scale (GCS) | Baseline up to Week 280
  PedsQL GCS is designed to measure health-related quality of life in pediatric participants and adolescents (2 to 18 years of age). It encompasses 4 dimensions of functioning (physical [8 items], emotional [5 items], social [5 items], school [3 items]). Age groups: Toddler (2-4 years), Young pediatric (5-7 years), Pediatric (8-12 years), and Teens (13-17 years). Depending on the participant's age, the questionnaire may be completed by parent/caregiver as appropriate. For the Toddler group, the PedsQL GCS consist of 21 items, using a 5-point Likert scale (0 to 4); for all other groups, the PedsQL GCS consist of 23 items, with a 3-point Likert scale (0, 2, 4) for the young pediatric, and a 5-point Likert scale for the pediatric and teens groups. Scores are transformed on a scale from 0 to 100 where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicate improved quality of life.
Population Pharmacokinetic (PK) Model Parameter Estimate: Maximum Plasma Concentration (Cmax) of Mitapivat | Weeks 2, 8, 12, and 16
Population PK Model Parameter Estimate: Area Under the Concentration-time Curve (AUC) Derived From Plasma Concentrations of Mitapivat | Weeks 2, 8, 12, and 16
Concentration at Steady State (Css) of Mitapivat | Week 16: 6 and 8 hours postdose
Trough Concentration (Ctrough) of Mitapivat | Week 8: ≤30 minutes predose; Week 12: ≤30 minutes predose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (19):
- United States (11):
  - Stanford Medicine, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Emory, Atlanta, Georgia
  - UChicago Medicine, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St Jude's Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Centre hospitalier Universitaire de Sainte-Justine, Montreal, Quebec, Canada
- Hôpital Pellegrin, Bordeaux, Aquitaine, France
- Germany (2):
  - Universitatsklinikum Wurzburg, Würzburg, Bavaria
  - Charite - UB - CVK - Medizinische Klinik, Berlin
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario Infantil Nino Jesus, Madrid
- CHUV University Hospital of Lausanne, Lausanne, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No